CLINICAL TRIAL: NCT05637086
Title: Clinical Study Evaluating and Comparing the Safety and the Possible Efficacy of Pentoxifylline and Celecoxib in Patients With Grand-Mal Epilepsy Treated by Phenytoin Monotherapy
Brief Title: Clinical Study Evaluating Safety of Pentoxifylline and Celecoxib in Patients With Grand-Mal Epilepsy Treated by Phenytoin Monotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Collaborators: Tanta University (Other); Principal Investigator Maha Ahmed Younis, PhD Pharmacy Practice Department- Horus University (Unknown)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22.09.108
Record Dates: First submitted 2022-11-27; First posted 2022-12-05 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Phenytoin; Pentoxifylline; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): This group will receive 100 mg of phenytoin 3 times daily for 6 months.
  Interventions: Drug: Phenytoin
- Pentoxifylline group (Active Comparator): This group will receive 100 mg of phenytoin 3 times daily plus pentoxifylline 400 mg two times daily for 6 months
  Interventions: Drug: Phenytoin; Drug: Pentoxifylline 400 MG
- Celecoxib group (Active Comparator): This group will receive 100 mg of phenytoin 3 times daily plus celecoxib 200 mg once daily for 6 months
  Interventions: Drug: Phenytoin; Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: Phenytoin — Phenytoin remains a highly effective anti-epileptic drug, especially in generalized seizure management. Unfortunately, phenytoin efficacy on epileptic seizure is apparently reduced with its chronic use
Drug: Pentoxifylline 400 MG — Pentoxifylline (PTX) has a well validated immune modulatory and anti-inflammatory efficacy
  Arms: Pentoxifylline group
Drug: Celecoxib 200mg — Celecoxib is a nonsteroidal anti-inflammatory drug (NSAID) used to treat mild to moderate pain and help relieve symptoms of arthritis
  Arms: Celecoxib group

SUMMARY:
Epilepsy is a chronic neurological disorder affecting millions of people all over the world. Epileptic seizures are caused by abnormal synchronized electrical neuronal discharges that could be either focal or widespread. Pathogenesis of epilepsy involves multiple processes including genetics, oxidative stress, ion channels, neuroinflammation, and cellular damage through autophagy and apoptosis.

Neuroinflammation is considered one of the most important factors contributing critically to epileptogenesis.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged ≥ 18 years old. Patients with grand mal epilepsy on phenytoin monotherapy. Women with a negative pregnancy test and women on effective contraception

Exclusion Criteria:

- Patients with significant liver and kidney function abnormalities. Alcohol and/or drug abusers. Patients with known allergies to the study medications Patients with known allergy to sulfonamides (cross hypersensitivity with celecoxib).

Pregnant women and women with a planned pregnancy. Subjects on medication are known to have possible positive effects on epilepsy. Patients who are currently using other antiepileptic drugs. Patients with CVD and a history of coronary artery bypass graft (CABG) surgery. Patients on aspirin or fluconazole therapy Patients with a recent retinal or cerebral hemorrhage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
The clinical outcome will be assessed through Quality of Life questionnaire (QOLIE-31) | 6 months
  Caregivers will complete the questionnaire for assessing the quality of life in epileptic patients.

SECONDARY OUTCOMES:
The secondary outcome is the change in the serum level of the measured biological parameters | 6 months
  The secondary outcome is the change in the serum level of the measured biological parameters such as High mobility group protein B1 (HMGB-1) serum level, and Nuclear Factor Kappa B (NF-κB) serum level

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Younis MA, El-Haggar SM, Mustafa W, Mostafa TM. Pentoxifylline as Adjuvant Therapy in Patients with Generalized Epilepsy Treated with Phenytoin: A Randomized Controlled Study. Mol Neurobiol. 2025 Dec;62(12):15978-15987. doi: 10.1007/s12035-025-05214-8. Epub 2025 Jul 30. PMID 40739381